CLINICAL TRIAL: NCT06759038
Title: Comparison Between C-MAC Blade D Video Laryngoscope and Macintosh Laryngoscope for Double Lumen Tube Insertion in Patients Undergoing Elective Thoracic Surgeries
Brief Title: C-MAC Blade D Video Vs Macintosh Laryngoscope for Double Lumen Tube Insertion
Acronym: DLT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shaheed Mohtarma Benazir Bhutto Institue of Trauma (Other)
Responsible Party: Principal Investigator, Sidra Tahir, Principal Investigator, Shaheed Mohtarma Benazir Bhutto Institue of Trauma
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: ERC-000146/SMBBIT/2024
Record Dates: First submitted 2024-12-11; First posted 2025-01-06 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2024-12

CONDITIONS: Video Laryngoscope; Double Lumen Tube Intubation; Elective Thoracic Surgery

STUDY DESIGN:
Intervention Model Description: There are two groups of participants Group A and Group B. Allocation of participants in each group is done by basic randomization.
Who Masked: Participant
Masking Description: Only participant is unaware that which type of intervention is using over him.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Video laryngoscope Group (Experimental): Those participants who will randomly assigned for intubations with C-MAC Blade D Video laryngoscope are placed in Group A
  Interventions: Device: C-MAC blade D video laryngoscope
- Macintosh laryngoscope Group (Active Comparator): Those participants who will randomly assigned for intubations with Macintosh Laryngoscope are placed in Group B
  Interventions: Device: Macintosh Laryngoscope

INTERVENTIONS:
Device: C-MAC blade D video laryngoscope — C-MAC blade D Video Laryngoscope is used for difficult intubation and for better glottic view
  Arms: Video laryngoscope Group
Device: Macintosh Laryngoscope — Macintosh Laryngoscope is conventional laryngoscope used generally for intubations
  Arms: Macintosh laryngoscope Group

SUMMARY:
The goal of this clinical trial is to know which type of laryngoscope is better for Double Lumen Tube (DLT) insertion, in participants undergoing elective thoracic surgeries.

The main question aim to answer is Is C-MAC blade D video laryngoscope better than Macintosh laryngoscope for DLT insertion in term of time taking for intubation and hemodynamic changes to laryngoscopy? Researchers are comparing two groups of participants

* Participants in Group A are receiving intubation from C-MAC blade D video laryngoscope.
* Participants in Group B are receiving intubations from Macintosh laryngoscope.

DETAILED DESCRIPTION:
Double Lumen Tube (DLT) is a common airway management device, used to implement lung isolation technique during thoracic surgeries. Intubation of DLT is challenging because it is much larger in diameter and rotational insertion technique is associated with significant risk of prolong intubation, intubation failure, greater hemodynamic changes and airway trauma.

Objective of this study is to compare the outcome C-MAC blade D video laryngoscope and Macintosh laryngoscope for DLT insertion, in term of time taking for DLT intubation and hemodynamic changes to laryngoscopy.

This study is conducting at Department of Anesthesiology at SMBBIT, Pakistan. Data is collecting after taking approval from Ethical Review Committee and written informed consent from participants.

Participants are enrolling by primary investigator, day before surgery. All participants are undergoing simple randomization by lottery method.

During induction of aesthesia, time for intubation is noting from introduction of the laryngoscope blade till three complete capnograph cycles.

Participants have also been assessed for hemodynamic parameters {Heart Rate (HR), Systolic Blood Pressure (SBP), Diastolic Blood Pressure (DBP) and Mean Arterial Pressure (MAP)} to intubation at 0 (Baseline), 1st Minute , 3rd Minute and 5th Minute after intubation.

After Completing data collection, Data analysis will be done by using SPSS version 26.

ELIGIBILITY:
Inclusion Criteria:

* Mallampati 1 and 2.
* ASA 1 and 2.
* Patients who will be prepared for elective thoracic surgeries under general anesthesia.

Exclusion Criteria:

* Pregnant Patients.
* Patients with anticipated difficult airway.
* Patients with limited neck extension.
* Thyromental distance less than 6.5cm.
* BMI greater than 35. (Weight in kilogram (kg) divided by height in meters squared)
* Patients at a risk of aspiration.
* Failure to intubate the patient after 3 attempts.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-12-03 (Actual); Primary Completion 2025-02-28 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Time for intubation | During induction of anesthesia, It will take 10 to 15 minutes
  1st outcome is time for intubation time for intubation will be noted during intubation of Double Lumen Tube. Time start from introduction of laryngoscope blade till three complete capnograph cycles.
Heart Rate changes to laryngoscopy | From enrollment till completion it will take approximately 24 hours
  Heart Rate of a patient will be noted before induction of Anaesthesia as baseline heart rate and will be labelled as 0. Then at 1 minute, at 3 minutes and at 5 minutes after intubation, and labelled as 1 ,3 & 5.
Blood pressure changes to laryngoscopy | Time from enrolment to completion will be 24 hours
  Changes of blood pressure to laryngoscopy as Systolic Blood Pressure (SBP), Diastolic Blood Pressure (DPB) and Mean Arterial Pressure (MAP) will be noted before induction of anesthesia as baseline and labelled as 0. Then at 1 minute, 3 minutes and 5 minutes after intubation and labelled as 1, 3 and 5.

CONTACTS AND LOCATIONS:
Locations (1):
- Shaheed Mohtarma Benazir Bhutto Institute of Trauma, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No
Patient Confidentiality: Sharing IPD could compromise patient confidentiality and anonymity Informed Consent: Participants are not providing informed consent for their data to be shared and it could raise ethical concerns.

REFERENCES:
- [Background] Smereka J, Ladny JR, Naylor A, Ruetzler K, Szarpak L. C-MAC compared with direct laryngoscopy for intubation in patients with cervical spine immobilization: A manikin trial. Am J Emerg Med. 2017 Aug;35(8):1142-1146. doi: 10.1016/j.ajem.2017.03.030. Epub 2017 Mar 16. PMID 28341185
- [Background] Kim YS, Song J, Lim BG, Lee IO, Won YJ. Different classes of videoscopes and direct laryngoscopes for double-lumen tube intubation in thoracic surgery: A systematic review and network meta-analysis. PLoS One. 2020 Aug 28;15(8):e0238060. doi: 10.1371/journal.pone.0238060. eCollection 2020. PMID 32857788
- [Background] Liu HH, Dong F, Liu JY, Wei JQ, Huang YK, Wang Y, Zhou T, Ma WH. The use of ETView endotracheal tube for surveillance after tube positioning in patients undergoing lobectomy, randomized trial. Medicine (Baltimore). 2018 Dec;97(49):e13170. doi: 10.1097/MD.0000000000013170. PMID 30544376
- [Background] Tao D, Zhang G, Zheng X, Wang X, Gao G, Yang Z, Lin Y, Lu L. Feasibility study of intubation in lateral position using Viva-sight double-lumen tube combined with video laryngoscope in patients undergoing pulmonary lobectomy. Asian J Surg. 2024 Jan;47(1):373-379. doi: 10.1016/j.asjsur.2023.08.199. Epub 2023 Sep 9. PMID 37696694